CLINICAL TRIAL: NCT04892797
Title: Understanding Immunology and Patient Outcomes of COVID-19: A 1-Year Longitudinal Follow-Up Study of Hospitalized Patients
Brief Title: Understanding Immunology and Patient Outcomes of COVID-19 in Hospitalized Patients
Status: Terminated | Type: Observational
Why Stopped: Grant application to fund this work was not funded. We won't be posting data for this study.
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Renee Stapleton, Professor of Medicine, University of Vermont
Other Study IDs: 00001369
Record Dates: First submitted 2021-02-09; First posted 2021-05-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19+: Hospitalized patients with Covid-19 infection confirmed by PCR test
  Interventions: Other: Covid-19+ observational

INTERVENTIONS:
Other: Covid-19+ observational — This is observational--there is no intervention

SUMMARY:
The adaptive immune response, consisting of antiviral T and B cells, is critical for providing protection against viruses such as SARS-CoV-2, both during an active infection and later following a subsequent exposure. They can both also potentially contribute to pathogenesis if they are overstimulated. Despite these advances in knowledge, there are still significant gaps in understanding of what constitutes a protective or immunopathologic immune response and its durability.

Significant knowledge gaps also remain pertaining to the early recognition of COVID patients with increased risk of clinical deterioration who require continued hospitalization and the use of more intensive treatments designed to improve outcomes. Data from non-COVID patients with MI show that platelet surface expression of FcγRIIa, the low-affinity receptor for the Fc fragment of immunoglobulin (Ig) G, identifies patients at high and low risk of subsequent cardiovascular events. Platelet expression of FcγRIIa is increased by interferon γ20 that is significantly elevated in severe COVID-19 infections. The high prevalence of arterial thrombosis among COVID-19 patients and the central role of thrombosis in respiratory failure support the hypothesis that elevated platelet expression of FcγRIIa will identify COVID patients at increased risk of thrombotic complications and clinical deterioration.

In addition to the potential role of platelet activation in thrombosis associated with COIVD-19, the endothelium may also play a significant role. The investigators hypothesize that elevated EMPs in plasma will identify patients at high risk of thrombosis and clinical deterioration.

To begin to address the knowledge gaps above and obtain preliminary data for future large grant submission, the investigators propose a small, prospective, single-center cohort study that will enroll patients hospitalized for COVID-19 infection and exhibiting a range of disease severity. Biosamples will be obtained and used to study T and B cells, antibody repertoire, and durability of protective immunity, and also to quantify platelet expression of FcγRIIa and circulating EMPs, as described in the protocol.

DETAILED DESCRIPTION:
Since December 2019, the novel coronavirus (SARS-CoV-2) and associated COVID-19 illness has spread worldwide. Globally, there are >86 million infections and over 1.8 million confirmed deaths, with the pandemic continuing at record levels throughout the USA. While new data on COVID-19 are emerging daily, several knowledge gaps remain, including understanding of the adaptive immune response to infection, the propensity for infected patients to experience thrombotic events, and identification of biomarkers that might predict clinical deterioration.

The adaptive immune response, consisting of antiviral T and B cells, is critical for providing protection against viruses such as SARS-CoV-2, both during an active infection and later following a subsequent exposure. They can both also potentially contribute to pathogenesis if they are overstimulated. Much has been learned about the T and B cell responses to SARS-CoV-2 since the beginning of the COVID-19 pandemic. The most comprehensive study to date shows that most individuals make a balanced T and B cell response that persists for at least 8 months. Despite these advances in knowledge, there are still significant gaps in understanding of what constitutes a protective or immunopathologic immune response and their durability.

Significant knowledge gaps also remain pertaining to the early recognition of COVID patients with increased risk of clinical deterioration who require continued hospitalization and the use of more intensive treatments designed to improve outcomes. In addition, the identification of low risk patients who can be discharged from the hospital would reduce the use of potentially scarce medical resources, particularly during a surge. Among patients with thrombosis, 49% required critical care and 43% died. Data from non-COVID patients with MI show that platelet surface expression of FcγRIIa, the low-affinity receptor for the Fc fragment of immunoglobulin (Ig) G, identifies patients at high and low risk of subsequent cardiovascular events. Platelet expression of FcγRIIa is increased by interferon γ20 that is significantly elevated in severe COVID-19 infections. Because FcγRIIa amplifies platelet activation, greater expression of FcγRIIa on the surface of the platelet increases platelet reactivity. The high prevalence of arterial thrombosis among COVID-19 patients and the central role of thrombosis in respiratory failure support the hypothesis that elevated platelet expression of FcγRIIa will identify COVID patients at increased risk of thrombotic complications and clinical deterioration.

In addition to the potential role of platelet activation in thrombosis associated with COIVD-19, the endothelium may also play a significant role. The endothelium is a key site of entry for COVID-19 infection and endothelial injury contributes to thrombotic events that increase morbidity and mortality. Endothelial microparticles (EMPs), submicron membranous vesicles indicating endothelial activation and injury, are released by the endothelium into blood and reflect the competency of endothelial function by identifying endothelial activation and injury, which promote thrombosis. Circulating EMPs can be quantified with the use of flow cytometry. The investigators hypothesize that elevated EMPs in plasma will identify patients at high risk of thrombosis and clinical deterioration.

To begin to address the knowledge gaps above and obtain preliminary data for future large grant submission, the investigators propose a small, prospective, single-center cohort study that will enroll patients hospitalized for COVID-19 infection and exhibiting a range of disease severity. Blood will be obtained on study days 1, 3±1, 7±1 (and every 7±1 days thereafter up to day 28 while hospitalized), and again at 12 months of follow up. Nasopharyngeal (NP) swabs will be collected on these same study days through day 28, but not at 12 months. These biosamples will be used to study T and B cells, antibody repertoire, and durability of protective immunity, and also to quantify platelet expression of FcγRIIa and circulating EMPs, as described in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) at the time of consent
2. Positive COVID-19 PCR test result

Exclusion Criteria:

1. Expected death or withdrawal of life-sustaining treatments within 3 days
2. Hemoglobin ≤7.0 at the time of consent
3. Unable to provide consent and no legally authorized representative (LAR) identified or reached by phone
4. Pregnant
5. Incarcerated
6. Physician declines patient enrollment (attending physician or study physician)
7. Patient or LAR do not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients hospitalized at the University of Vermont Medical Center who have a positive test result for COVID-19. These patients are expected to have a greater acuity of illness and burden of disease based on the fact that they require inpatient care. Enrolling hospitalized patients ensures a greater opportunity to collect serial biological specimens over the course of the illness due to the proximity of the patient to medical and research staff and UVM laboratories.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the polyfunctionality and frequency of antiviral CD4 and CD8 T cells. | Four weeks (while hospitalized)
  The investigators hypothesize patients with severe disease will have higher frequencies of antiviral T cells that contribute to the cytokine storm observed in the most severe cases of COVID-19.
To compare the polyfunctionality and frequency of antiviral CD4 and CD8 T cells. | 12 months after hospital admission
  The investigators hypothesize patients with severe disease will have higher frequencies of antiviral T cells that contribute to the cytokine storm observed in the most severe cases of COVID-19.
To compare the frequency of plasmablasts (early B cells that produce antiviral antibodies) and plasma antiviral antibody titer during acute infection. | Four weeks (while hospitalized)
  The investigators predict that patients with severe disease will have greater numbers of antiviral plasmablasts and plasma antiviral antibody levels compared to those with mild disease.
To compare the frequency of plasmablasts (early B cells that produce antiviral antibodies) and plasma antiviral antibody titer during acute infection. | 12 months after hospital admission
  The investigators predict that patients with severe disease will have greater numbers of antiviral plasmablasts and plasma antiviral antibody levels compared to those with mild disease.
The number of virus specific CD4 T cells will be measured using flow cytometry. | Four weeks (while hospitalized)
  The investigators hypothesize that severe disease will result in the formation of higher magnitude antiviral B and T cell CHRMS (Medical) #STUDY00001369 Approved: 1/25/2021 4Human subjects protocol form 7/19/19responses during acute disease due to increased viral load and antigen in these patients. The investigators further predict that higher frequency T and B cells during acute disease will correlate with more robust durability of these responses during convalescence.
The number of virus specific CD8 T cells will be measured using flow cytometry. | Four weeks (while hospitalized)
  The investigators hypothesize that severe disease will result in the formation of higher magnitude antiviral B and T cell CHRMS (Medical) #STUDY00001369 Approved: 1/25/2021 4Human subjects protocol form 7/19/19responses during acute disease due to increased viral load and antigen in these patients. The investigators further predict that higher frequency T and B cells during acute disease will correlate with more robust durability of these responses during convalescence.
The number of virus specific CD4 T cells will be measured using flow cytometry. | 12 months after hospital admission
  The investigators hypothesize that severe disease will result in the formation of higher magnitude antiviral B and T cell CHRMS (Medical) #STUDY00001369 Approved: 1/25/2021 4 Human subjects protocol form 7/19/19 responses during acute disease due to increased viral load and antigen in these patients. The investigators further predict that higher frequency T and B cells during acute disease will correlate with more robust durability of these responses during convalescence.
The number of virus specific CD8 T cells will be measured using flow cytometry. | 12 months after hospital admission
  The investigators hypothesize that severe disease will result in the formation of higher magnitude antiviral B and T cell CHRMS (Medical) #STUDY00001369 Approved: 1/25/2021 4Human subjects protocol form 7/19/19responses during acute disease due to increased viral load and antigen in these patients. The investigators further predict that higher frequency T and B cells during acute disease will correlate with more robust durability of these responses during convalescence.
To obtain preliminary data on platelet activation in patients hospitalized with COVID-19 | Four weeks (while hospitalized)
  To compare platelet activation, measured by platelet surface FcγRIIa while in hospital and 12 months after infection, in patients with severe (i.e., mechanical ventilation in ICU) vs. non-severe (hospitalized, but not in an ICU) COVID-19 disease.
To obtain preliminary data on platelet activation in patients hospitalized with COVID-19 | 12 months after hospital admission
  To compare platelet activation, measured by platelet surface FcγRIIa while in hospital and 12 months after infection, in patients with severe (i.e., mechanical ventilation in ICU) vs. non-severe (hospitalized, but not in an ICU) COVID-19 disease.
To obtain preliminary data on endothelial activation in patients hospitalized with COVID-19 | Four weeks (while hospitalized)
  To compare endothelial activation, measured by circulating EMPs while in hospital and 12 months after infection, in patients with severe (i.e., mechanical ventilation in ICU) vs. non-severe (hospitalized, but not in an ICU) COVID-19 disease.
To obtain preliminary data on endothelial activation in patients hospitalized with COVID-19 | 12 months after hospital admission
  To compare endothelial activation, measured by circulating EMPs while in hospital and 12 months after infection, in patients with severe (i.e., mechanical ventilation in ICU) vs. non-severe (hospitalized, but not in an ICU) COVID-19 disease.
Preliminarily determine if the FcγRIIa and EMPs have utility as biomarkers | Four weeks (while hospitalized)
  To preliminarily determine if the FcγRIIa and EMPs have utility as biomarkers for prediction of thrombotic events and clinical deterioration in hospitalized patients with COVID-19.
Preliminarily determine if the FcγRIIa and EMPs have utility as biomarkers | 12 months after hospital admission
  To preliminarily determine if the FcγRIIa and EMPs have utility as biomarkers for prediction of thrombotic events and clinical deterioration in hospitalized patients with COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Stapleton, MD, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided